CLINICAL TRIAL: NCT02692768
Title: The Effect of Music Therapy Intervention on Pain and Anxiety in Adult Patients Undergoing Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: April Armstrong (Other)
Responsible Party: Sponsor-Investigator, April Armstrong, Principal Investigator / Sponsor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004093
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Arthritis
Keywords: total shoulder arthroplasty; total shoulder replacement; adult; reverse shoulder arthroplasty
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Music Therapy (Active Comparator): Live sedative guitar playing within a limited chord progression will be utilized. Added to this music will be vocal and verbal therapeutic suggestion for active listening, focused breathing, muscle relaxation, and guided imagery. Patients will choose from one of three nature scene options for the guided imagery in order to include patient preference of content. This treatment group will experience this music intervention live, including patient-centered interaction with the music therapist and education for repeated use of the routine on recording.
  Interventions: Other: Live Music Therapy
- Recorded Music Therapy (Active Comparator): Recorded sedative guitar playing within a limited chord progression will be utilized. Added to this music will be vocal and verbal therapeutic suggestion for active listening, focused breathing, muscle relaxation, and guided imagery. Patients will choose from one of three nature scene options for the guided imagery in order to include patient preference of content. This treatment group will be given a recording of their chosen music relaxation routine for use throughout the study process.
  Interventions: Other: Recorded Music Therapy
- Control (Active Comparator): This group will receive standard of care with no music therapy intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Live Music Therapy — Patients in this arm will meet with the music therapist to indicate preferences for one of three guided imagery scenarios to be included in their music-assisted relaxation routine. Patients will then receive live music relaxation and education for practice using a CD. Once admitted for surgery, patients will be seen immediately prior to going to the OR in the SDU, immediately following surgery in the PACU, and then within 12-24 hours of surgery on the inpatient floor. Pain and anxiety measures will be gathered at routine follow-up appointments following discharge (2 weeks and 6 months post-operatively).
  Arms: Live Music Therapy
Other: Recorded Music Therapy — Patients in this arm will meet with the music therapist to indicate preferences for one of three guided imagery scenarios to be included in their music-assisted relaxation routine. Patients will then receive explanation for using the recorded routine on CD. Once admitted for surgery, patients will be seen immediately prior to going to the OR in the SDU, immediately following surgery in the PACU, and then within 12-24 hours of surgery on the inpatient floor. Pain and anxiety measures will be gathered at routine follow-up appointments following discharge (2 weeks and 6 months post-operatively).
  Arms: Recorded Music Therapy
Other: Control — Patients will receive standard of care without any music therapy intervention. These patients will have pain and anxiety measures taken at the same contact points as the music therapy intervention groups.
  Arms: Control

SUMMARY:
The purpose of this study is to determine if music therapy interventions as adjunct to standard surgical care reduces pre- and post-operative pain and anxiety in patients undergoing total shoulder arthroplasty as compared with patients who receive standard of care without music therapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded clinical trial. The primary objective is to measure differences in pain and anxiety scores before and after music therapy interventions as compared to patients who do not receive music therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Body mass: 50-125 kg (inclusive )
* Elective total or reverse total shoulder arthroplasty surgery by the study investigator
* Gender: male or female (non-pregnant)
* American Society of Anesthesiologists physical classification scale 1-3
* Fluent in written and spoken English
* Patients capable of giving informed consent

Exclusion Criteria:

* Age less than 18 years of age
* Non-elective surgery by the study investigator
* Pregnancy
* American Society of Anesthesiologists physical classification scale 4-5
* Non-English speaking persons
* Diagnosis of cognitive disorder or musicogenic epilepsy
* Pre-existing hearing problems, defined as inability to independently hear speech or music at average volume
* Diagnosis of cognitive disorder including psychosis and dementia and/or musicogenic epilepsy
* Anatomical abnormalities of the shoulder such as cancerous lesions or congenital defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain scores on the visual analog scale at 6 months | 6 months
  Patients will be asked to return to the research site a total of six times (pre-operative, pre-surgery, post-surgery, recovery visit (12-24 hours after surgery), two-weeks post-operative visit, and 6 months post-operative visit). Pain scores will be recorded at each of these times.

SECONDARY OUTCOMES:
Change from baseline in anxiety scores on the PROMIS Emotional Distress-Anxiety-Short Form at 6 months | 6 months
  Patients will be asked to return to the research site a total of six times (pre-operative, pre-surgery, post-surgery, recovery visit (12-24 hours after surgery), two-weeks post-operative visit, and 6 months post-operative visit). Anxiety scores will be recorded at each of these times.

CONTACTS AND LOCATIONS:
Overall Officials: April D Armstrong, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy JC, Everding NG, Gil CC Jr, Stephens S, Giveans MR. Speed of recovery after shoulder arthroplasty: a comparison of reverse and anatomic total shoulder arthroplasty. J Shoulder Elbow Surg. 2014 Dec;23(12):1872-1881. doi: 10.1016/j.jse.2014.04.014. Epub 2014 Jun 26. PMID 24981553
- [Background] The Joint Commission. (2015). Facts about pain management. Retrieved from http://www.jointcommicssion.org/pain_management on 09.08.2015.
- [Background] The Joint Commission. (2014). Clarification of the pain management standard. Joint Commission Perspectives, 34, 11, 11.
- [Background] Epker J, Block AR. Presurgical psychological screening in back pain patients: a review. Clin J Pain. 2001 Sep;17(3):200-5. doi: 10.1097/00002508-200109000-00003. PMID 11587109
- [Background] Rafer L, Austin F, Frey J, Mulvey C, Vaida S, Prozesky J. Effects of jazz on postoperative pain and stress in patients undergoing elective hysterectomy. Adv Mind Body Med. 2015 Winter;29(1):6-11. PMID 25607117
- [Background] Dileo, C., Bradt, J. (2005). Medical music therapy: a meta-analysis & agenda for future research. Cherry Hill, NJ: Jeffrey Books.
- [Background] Cepeda MS, Carr DB, Lau J, Alvarez H. WITHDRAWN: Music for pain relief. Cochrane Database Syst Rev. 2013 Oct 25;2013(10):CD004843. doi: 10.1002/14651858.CD004843.pub3. PMID 24163271
- [Background] What is music therapy? Retrieved from http://www.musictherapy.org/about/musictherapy/
- [Background] Tan X, Yowler CJ, Super DM, Fratianne RB. The Interplay of Preference, Familiarity and Psychophysical Properties in Defining Relaxation Music. J Music Ther. 2012 Summer;49(2):150-79. doi: 10.1093/jmt/49.2.150. PMID 26753216
- [Background] Robb, S., Nichols, R., Rutan, R., Bishop, B., & Parker, J. (1995). The effects of music assisted relaxation on perioperative anxiety. Journal of Music Therapy, 32, 2-21.
- [Background] Stouffer JW, Shirk BJ, Polomano RC. Practice guidelines for music interventions with hospitalized pediatric patients. J Pediatr Nurs. 2007 Dec;22(6):448-56. doi: 10.1016/j.pedn.2007.04.011. PMID 18036465
- [Background] Modesti PA, Ferrari A, Bazzini C, Costanzo G, Simonetti I, Taddei S, Biggeri A, Parati G, Gensini GF, Sirigatti S. Psychological predictors of the antihypertensive effects of music-guided slow breathing. J Hypertens. 2010 May;28(5):1097-103. doi: 10.1097/HJH.0b013e3283362762. PMID 20160655
- [Background] Madson AT, Silverman MJ. The effect of music therapy on relaxation, anxiety, pain perception, and nausea in adult solid organ transplant patients. J Music Ther. 2010 Fall;47(3):220-32. doi: 10.1093/jmt/47.3.220. PMID 21275333
- [Background] Kleiber C, Adamek MS. Adolescents' perceptions of music therapy following spinal fusion surgery. J Clin Nurs. 2013 Feb;22(3-4):414-22. doi: 10.1111/j.1365-2702.2012.04248.x. Epub 2012 Sep 18. PMID 22985428
- [Background] Chi GC, Young A. Selection of music for inducing relaxation and alleviating pain: literature review. Holist Nurs Pract. 2011 May-Jun;25(3):127-35. doi: 10.1097/HNP.0b013e3182157c64. PMID 21508712
- [Background] Bradt, J. (2010). The effects of music entrainment on postoperative pain perception in pediatric patients. Music and medicine, 2(3):150-57.
- [Background] Mitchell LA, MacDonald RA. An experimental investigation of the effects of preferred and relaxing music listening on pain perception. J Music Ther. 2006 Winter;43(4):295-316. doi: 10.1093/jmt/43.4.295. PMID 17348757
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Cohen J. (1988) Statistical Power Analysis for the Behavioral Sciences (2nd ed). Lawrence Erlbaum Associates, Publisher